CLINICAL TRIAL: NCT02735642
Title: High-yield HIV Testing, Facilitated Linkage to Care, and Prevention for Female Youth in Kenya (GIRLS)
Brief Title: High-yield HIV Testing, Facilitated Linkage to Care, and Prevention for Female Youth in Kenya
Acronym: GIRLS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: Kenyatta National Hospital (Other Government); Impact Research & Development Organization (Other); National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Supportive Care
Other Study IDs: 1512016985; 1R01AI122797 (NIH)
Record Dates: First submitted 2016-03-29; First posted 2016-04-13 (Estimated); Results first posted 2020-11-02 (Actual); Last update posted 2021-11-02 (Actual); Status verified 2021-10

CONDITIONS: HIV; Adolescent Behavior
MeSH Terms: conditions — Adolescent Behavior | interventions — Spermine Synthase

STUDY DESIGN:
Intervention Model Description: Adaptive linkage to care interventions for newly diagnosed HIV-positive participants. Total N recruited will depend on HIV prevalence found in the study.
Who Masked: Participant
Masking Description: We utilized an approach called permuted blocks randomization for participant assignment to the SMART trial linkage to care intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- SMART Randomization 1 - Referral (Experimental): Participants who are HIV positive will be enrolled in the SMART trial adaptive linkage to care intervention pilot. (HIV Positive Cohort approximately N=108).
  Interventions: Behavioral: SMART Randomization 1 - Referral
- SMART Randomization 1 - Referral and SMS (Experimental): Participants who are HIV positive will be enrolled in the SMART trial adaptive linkage to care intervention pilot. (HIV Positive Cohort approximately N=108).
  Interventions: Behavioral: SMART Randomization 1 - Referral and SMS
- SMART Randomization 2 - SMS (Experimental): HIV positives that have not successfully linked to care after the first randomization will be re-randomized to receive either an SMS message or economic incentive to link to care. (HIV Positive Cohort approximately N=108).
  Interventions: Behavioral: SMART Randomization 2 - SMS
- SMART Randomization 2 - Incentive (Experimental): HIV positives that have not successfully linked to care after the first randomization will be re-randomized to receive either an SMS message or economic incentive to link to care. (HIV Positive Cohort approximately N=108).
  Interventions: Behavioral: SMART Randomization 2 - Incentive
- High Risk Negative Cohort (N=185) (Other): A subset of negatives identified as 'high risk' from the CAPI baseline survey will be invited to participate in the primary prevention intervention (N=185).
  Interventions: Behavioral: High Risk Negative Cohort (N=185)
- All participants. Approximately (N=1200) (Other): HIV testing options that female youth can choose from include: (1) oral fluid HIV self-testing (OHIVST) at their convenience; (2) immediate staff-aided testing at home/mobile site; and (3) a referral to a health care facility where HIV testing will be done by a health care provider (standard facility-based HTS).
  Interventions: Other: All participants. Approximately (N=1200)

INTERVENTIONS:
Behavioral: SMART Randomization 1 - Referral — Participants will be randomized to receive standard referral to link to HIV care. When successfully linked to care, they will receive SMS reminders combined with health status surveys at 3, 6, 9, and 12 months. All participants will have viral loads and CD4 collected at baseline and at 12 months, viral loads collected again and an exit interview completed.
  Arms: SMART Randomization 1 - Referral
Behavioral: SMART Randomization 1 - Referral and SMS — Participants will be randomized to receive referral plus SMS to link to HIV care. When successfully linked to care, they will receive SMS reminders combined with health status surveys at 3, 6, 9, and 12 months. All participants will have viral loads and CD4 collected at baseline and at 12 months, viral loads collected again and an exit interview completed.
  Arms: SMART Randomization 1 - Referral and SMS
Behavioral: SMART Randomization 2 - SMS — Those that have not linked to care after the first randomization, will be re-randomized to receive an SMS message. When successfully linked to care, they will receive SMS reminders combined with health status surveys at 3, 6, 9, and 12 months. All participants will have viral loads and CD4 collected at baseline and at 12 months, viral loads collected again and an exit interview completed.
  Arms: SMART Randomization 2 - SMS
Behavioral: SMART Randomization 2 - Incentive — Those that have not linked to care after the first randomization, will be re-randomized to receive a one-time economic incentive. When successfully linked to care, they will receive SMS reminders combined with health status surveys at 3, 6, 9, and 12 months. All participants will have viral loads and CD4 collected at baseline and at 12 months, viral loads collected again and an exit interview completed.
  Arms: SMART Randomization 2 - Incentive
Behavioral: High Risk Negative Cohort (N=185) — A subset of negatives identified as 'high risk' from the CAPI baseline survey will be invited to participate in the primary prevention intervention (N=185). They will receive an SMS health promotion message with survey at 6 and 12 months. At 12 months, they will be re-tested for HIV and an exit interview completed.
  Arms: High Risk Negative Cohort (N=185)
Other: All participants. Approximately (N=1200) — HIV testing approaches that females can choose from include: (1) oral fluid HIV self-testing (OHIVST) at their convenience; (2) immediate staff-aided testing at home/mobile site; and (3) a referral to a health care facility where HIV testing will be done by a health care provider (standard facility-based HTS).
  All participants will receive a behavioral CAPI survey at baseline visit, an SMS HIV test experience satisfaction survey, and for those who choose the self-testing option, a staff-administered questionnaire.
  Arms: All participants. Approximately (N=1200)

SUMMARY:
Knowledge of HIV status is a first step towards accessing HIV care, treatment, and prevention services.The GIRLS study will rigorously compare two 'seek' recruitment strategies, three 'test' strategies, and two enhancements to an adaptive (SMART trial design) 'linkage' to care intervention, among young at-risk women, 15-24 years old, in Homa Bay County, western Kenya. Additionally, we will evaluate a scalable primary prevention messaging intervention to support identified HIV-negative young women in reducing HIV risk and adhering to recommended HIV re-testing recommendations. We will also conduct an economic evaluation, using cost effectiveness analyses to determine the relative utility of each seek, test, link, and prevention interventions.

Lessons learned will inform Government of Kenya, and other key policymakers, implementing partners and agencies throughout sub-Saharan Africa that are exploring policies about appropriate scale up of these multiple seek, test, link, retain, and prevention strategies to realize the dream of an AIDS-free future for adolescent girls and young women.

DETAILED DESCRIPTION:
The GIRLS study will inform best practices to increase adolescent girls and young women's uptake of HIV prevention, testing, and linkage for HIV to care services in a high-HIV burden African setting to optimize engagement in both the HIV prevention and care continua.

Aim 1: To determine the preferred recruitment venue and testing modality that targets and finds the highest number of HIV infected and at risk female youth aged 15-24 years in Homa Bay County, Nyanza region, western Kenya.

* This will be determined by examining the uptake and yield of previously undiagnosed HIV infection of the two (2) 'seek' strategies (community or home-based) and the three (3) 'test' strategies (self-testing, HIV testing services (HTS) in a home/mobile setting, or facility-based HTS) among female youth;

Aim 2: (a) To pilot and evaluate an adaptive intervention to link newly diagnosed HIV-positive female youth to treatment and care services; and (b) To identify barriers and facilitators to seeking HIV care services after receiving a positive diagnosis; (c) To identify barriers and facilitators to seeking HIV prevention services for high risk female youth after receiving a negative HIV test result; (d) To provide an HIV prevention intervention to a randomly selected subset of high risk negatives, and to re-test them; and

Aim 3: To conduct an economic evaluation, using cost effectiveness analyses to determine the relative utility of each seek, test, link, and prevention intervention.

ELIGIBILITY:
Inclusion Criteria:

* Able to understand spoken English or Kiswahili or Dholuo
* Resides in Homa Bay County
* Not previously diagnosed as HIV positive
* Willing to give informed consent or if younger than 18 years of age has a parent or guardian willing to provide consent in addition to the minor's assent

Exclusion Criteria:

* Male
* Unable to understand spoken English, or Kiswahili or Dholuo
* Females who do not meet age inclusion criteria
* Resides outside of Homa Bay County
* HIV positive
* If under 18 and not an emancipated minor, unable to get parental consent

Ages: 15 Years to 24 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 1198 (Actual)
Dates: Start 2017-05-15 (Actual); Primary Completion 2018-04-10 (Actual); Study Completion 2019-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ann E. Kurth, PhD, CNM, Principal Investigator — Yale University School of Nursing; Irene Inwani, MD, MPH, Principal Investigator — Kenyatta National Hospital; Kawango Agot, PhD, MPH, Principal Investigator — Impact Research & Development Organization
Locations (1):
- Impact Research & Development Organization, Kisumu, Kenya

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Inwani I, Chhun N, Agot K, Cleland CM, Buttolph J, Thirumurthy H, Kurth AE. High-Yield HIV Testing, Facilitated Linkage to Care, and Prevention for Female Youth in Kenya (GIRLS Study): Implementation Science Protocol for a Priority Population. JMIR Res Protoc. 2017 Dec 13;6(12):e179. doi: 10.2196/resprot.8200. PMID 29237583
- [Result] Inwani I, Chhun N, Agot K, Cleland CM, Rao SO, Nduati R, Kinuthia J, Kurth AE. Preferred HIV Testing Modalities Among Adolescent Girls and Young Women in Kenya. J Adolesc Health. 2021 Mar;68(3):497-507. doi: 10.1016/j.jadohealth.2020.07.007. Epub 2020 Aug 11. PMID 32792256

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled between May 2017 and April 2018 from three sites in Homa Bay County, Nyanza region, western Kenya. In fulfillment of Aim 1, we explored two recruitment approaches (homebased vs. mobile-event based) and three HIV testing options (oral self-test, staff-administered, or referral to health facility).
Pre-assignment Details: After participants completed HIV testing, only newly diagnosed participants living with HIV were enrolled into the SMART trial component of the study. This occurred from June 2017 to June 2018. Please note these are not additional participants, they are part of the N=1198 enrolled in the overall study.
Groups:
- Aim 1: Home-based Recruitment Strategy: In fulfillment of Aim 1, we explored the home-based recruitment approach and three HIV testing options (oral self-test, staff-administered, or referral to health facility), to see which recruitment approach and testing modality would yield the highest number of newly diagnosed adolescent girls and young women living with HIV.
- Aim 1: Mobile Event Based Recruitment Strategy: In fulfillment of Aim 1, we explored the mobile event based recruitment approach and three HIV testing options (oral self-test, staff-administered, or referral to health facility), to see which recruitment approach and testing modality would yield the highest number of newly diagnosed adolescent girls and young women living with HIV.
Period: Overall Study
Arm/Group | Aim 1: Home-based Recruitment Strategy | Aim 1: Mobile Event Based Recruitment Strategy
Started | 1046 | 152
Completed | 1046 | 152
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: This section summarizes the baseline characteristics of our study participants. Therefore N=1198.
Groups:
- Home-based Recruitment Strategy; Mobile Event Based Recruitment Strategy: We explored two recruitment approaches (homebased vs. mobile-event based) and three HIV testing options (oral self-test, staff-administered, or referral to health facility).
- Total: Total of all reporting groups
Arm/Group | Home-based Recruitment Strategy | Mobile Event Based Recruitment Strategy | Total
Number analyzed (Participants) | 1046 | 152 | 1198
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 20 [18 to 22] | 19 [18 to 22] | 20 [18 to 22]
Sex/Gender, Customized [Count of Participants; unit: Participants] — The number of adolescents and young women (AGYW) enrolled via each recruitment strategy. This study only enrolls AGYW.
  Participants
    Adolescent girls and young women | 1046 | 152 | 1198
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1046 | 152 | 1198
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Kenya | 1046 | 152 | 1198

OUTCOME MEASURES:

1. Primary Outcome: Number of Newly Diagnosed Adolescent Girls and Young Women Living With HIV
Description: Our primary outcome for comparisons of recruitment and testing strategies was the number of newly diagnosed adolescent girls and young women living with HIV.
Time Frame: Baseline
Measure: Count of Participants; unit: Participants
Groups:
- Home-based Recruitment Strategy: In fulfillment of Aim 1, we explored the home-based recruitment approach and three HIV testing options (oral self-test, staff-administered, or referral to health facility), to see which recruitment approach and testing modality would yield the highest number of newly diagnosed adolescent girls and young women living with HIV.
- Mobile Event Based Recruitment Strategy: In fulfillment of Aim 1, we explored the mobile event based recruitment approach and three HIV testing options (oral self-test, staff-administered, or referral to health facility), to see which recruitment approach and testing modality would yield the highest number of newly diagnosed adolescent girls and young women living with HIV.
Arm/Group | Home-based Recruitment Strategy | Mobile Event Based Recruitment Strategy
Number analyzed (Participants) | 1046 | 152
Participants | 23 | 9

2. Secondary Outcome: SMART Trial Pilot to Link Newly Diagnosed Adolescent Girls and Young Women to HIV Care Services.
Description: After completing HIV testing, newly diagnosed adolescent girls and young women (AGYW) (N=32) participated in an adaptive intervention pilot to figure out the best way to support those newly diagnosed with HIV with initial linkage to care. The SMART trial pilot consisted of two randomizations. In the first randomization, AGYW were assigned to either standard referral (counseling and a referral note) or standard referral plus SMS message; those not linked to care after the first randomization (within a 2-week period) were randomized a second time to receive either a SMS message or financial incentive to link to care.
Time Frame: Baseline to about 6 weeks
Population: Please note our SMART trial is underpowered because HIV prevalence was lower than expected. In the outcome measure data table below, we report the total numbers allocated to each intervention and the number of participants who successfully linked to care.
Measure: Count of Participants; unit: Participants
Groups:
- SMART Randomization 1 - Referral: Newly diagnosed adolescent girls and young women living with HIV were enrolled into a SMART trial to pilot adaptive interventions to support them with initial linkage to treatment and care services.
  In the first randomization, participants in this arm were randomized to referral.
- SMART Randomization 1 - Referral and SMS: Newly diagnosed adolescent girls and young women living with HIV were enrolled into a SMART trial to pilot adaptive interventions to support them with initial linkage to treatment and care services.
  In the first randomization, participants in this arm were randomized to receive referral and SMS message.
- SMART Randomization 2 - SMS: Newly diagnosed adolescent girls and young women living with HIV that have not successfully linked to care after the first randomization were re-randomized to receive either an SMS message or economic incentive to link to care.
  In this second randomization, participants in this arm were randomized to receive an SMS message.
- SMART Randomization 2 - Incentive: Newly diagnosed adolescent girls and young women living with HIV that have not successfully linked to care after the first randomization were re-randomized to receive either an SMS message or economic incentive to link to care.
  In this second randomization, participants in this arm were randomized to receive an economic incentive.
Arm/Group | SMART Randomization 1 - Referral | SMART Randomization 1 - Referral and SMS | SMART Randomization 2 - SMS | SMART Randomization 2 - Incentive
Number analyzed (Participants) | 15 | 17 | 1 | 1
Participants | 10 | 10 | 0 | 1

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the date of first participant enrollment, until the date the last participant completed follow-up (about one year for those who participated in the longitudinal follow-up).
Arm/Group | Home-based Recruitment Strategy | Mobile Event Based Recruitment Strategy
All-Cause Mortality (participants affected / at risk) | 0/1046 | 0/152
Serious Adverse Events (participants affected / at risk) | 0/1046 | 0/152
Other Adverse Events (participants affected / at risk) | 1/1046 | 1/152
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Home-based Recruitment Strategy (N=1046) | Mobile Event Based Recruitment Strategy (N=152)
Social Harms (Social circumstances) | 1 (1) | 1 (1) — Social harms are non-medical adverse events that may occur because of being in the study. Socials harms include difficulties in personal relationships, discrimination or stigma from the community or a family members as a result of study participation

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-09-09): https://cdn.clinicaltrials.gov/large-docs/42/NCT02735642/Prot_SAP_000.pdf